CLINICAL TRIAL: NCT01730248
Title: A Phase Ib, Open-label, Multi-center, Two-arm, Dose-finding Study to Assess Safety and Efficacy of the Oral Combination or INC424 (INC424) and BKM120 in Patients With Primary Myelofibrosis (PMF), Postpolycythemia Vera-myelofibrosis (PPV-MF), or Post-essential Thrombocythemia-myelofibrosis (PET-MF)
Brief Title: A Study to Find the Maximum Tolerated Dose of the Experimental Combination of the Drugs INC424 and BKM120 in Patients With Primary or Secondary Myelofibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision by Sponsor to to terminate the study early.
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC424A2104
Record Dates: First submitted 2012-11-12; First posted 2012-11-21 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2019-03

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis,; PMF,; PPV-MF,; PET-MF,; Primary Myelofibrosis,; Post-polycythemia vera myelofibrosis,; Post-essential thrombocythemia myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JAK Inhibitor Naive (Experimental): Two treatment periods applicable to all patients; Treatment Period (6 cycles / 28 days per cycle) and Extension Period ( 6 or more cycles of 28 days, with visits every 28days for 6 cycles and then visits every 12 weeks) following the treatment period dependent on patient continued eligibility. Two Study Phases: Dose Escalation Phase to determine maximum tolerated dose (MTD) / Recommended Phase II dose (RPIID) & an Expansion Phase
  Interventions: Drug: INC424; Drug: BKM120
- Prior JAK Inhibitor (Experimental): Two treatment periods applicable to all patients; Treatment Period (6 cycles / 28 days per cycle) and Extension Period (6 or more cycles of 28 days, with visits every 28 days for 6 cycles then visits every 12 weeks) following the treatment period dependent on patient continued eligibility. Two Study Phases: Dose Escalation Phase to determine MTD / RPIID & an Expansion Phase
  Interventions: Drug: INC424; Drug: BKM120

INTERVENTIONS:
Drug: INC424 — 5 mg tablets administered orally twice daily
Drug: BKM120 — 10 mg and 50 mg hard gelatin capsules administered orally once daily

SUMMARY:
The purpose of this phase Ib clinical trial is to evaluate the safety of the combination of INC424 and BKM120 in the myelofibrosis population and to establish the maximum tolerated dose and or the Recommended Phase II dose of the combination guided by the Bayesian dose escalation model. INC424 has shown efficacy in myelofibrosis (MF) and is approved in the US and EU for the treatment of MF. BKM120 is a PI3K inhibitor. Preclinical and early clinical experience support inhibition of the PI3K/mTOR pathway in MF as aberrant activation of the pathway has been observed in MF models and may contribute to the pathogenesis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PMF, PPV-MF or PET-MF irrespective of JAK2 mutation status
* Myelofibrosis patients requiring therapy must be classified as intermediate risk level 1 )1 or more prognostic factors defined by IWG) with at least one criteria other than age
* Must have palpable spleen of at least 5 cm from the costal margin to the point of greatest splenic profusion at Screening
* Must have active symptoms of MF (one symptom score of at least 5 or two symptom scores of at least 3 at Screening) (per MFSSF 0-10)
* PLT counts > or = 75X 10^9/L at Screening or Cycle 1 Day 1 (not with aid of transfusions

Exclusion Criteria:

* Pregnant or nursing women
* WOCBP not using highly effective methods of contraception
* Sexually active males who refuse condom use
* Previous Treatment with one of the following: PI3 K inhibitors and AKT inhibitors; JAK inhibitors that resulted in clinically significant toxicities per the Investigator;
* Patients who have had splenic irradiation within 12 months prior to Screening
* Patients with specific mood disorders
* Any history of bleeding diathesis
* Patients receiving the following treatments / medications:

EIAED within 2 wks. prior to study treatment; medication known to prolong QT interval or induce Torsades de Pointes; treatment with potent systemic systemic inhibitor or systemic inducer of CYP3A4; any use of drug that interferes with coagulation or inhibits PLT function

-current and willing candidates for a stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | baseline, when the maximum tolerated dose is established.
  The incidence of dose limiting toxicities will be analyzed to establish the maximum tolerated dose. To assess the maximum tolerated dose, labs and adverse events are monitored.

SECONDARY OUTCOMES:
Frequency of adverse events | after each cohort is enrolled at baseline until the maximum tolerated dose is established
  Adverse Events are monitored at each study visit and 30 days post last dose of study drug
Frequency of serious adverse events | after each cohort is enrolled at baseline until the maximum tolerated dose is established
  Serious Adverse events monitored at each study visit and 30 days post last dose of study drug
Abnormalities in vital signs | baseline, days 2, 8, 15, 22 of cycle 1, day 1 and 15 at Cycle 2, Day 1 from cycle 3 to 12, day 28 on Cycle 12 and every 12 weeks from Week 60 to 96 and at End of treatment
  cycle = 28 days
Laboratory test values including Imaging (electrocardiograms (ECGs), abdominal MRI/CT, ECHO/MUGA | Day 1, 2, 5, 8, 11, 18, 22, 25 of cycle 1, weekly in cycle 2, then at every scheduled visit including End of treatment visit
  ECGs are performed baseline, days 2, 8, 15, 22 of cycle 1 then day 1 from Cycle 2 to cycle 12, and at cycle 12 day 28 and every 12 weeks and end of treatment. Magnetic resonance imaging (MRI) or Cat Scan (CT) performed at baseline, cycle 4 day 1, cycle 7 day 1, cycle 12 day 28, then every 24 weeks , and end of treatment if not done in past 12 weeks. Echocardiography (ECHO) or Multiple Gated Acquisition (MUGA) is performed at baseline and then every 4 cycles until cycle 12, then every 24 weeks therafter or as clinically indicated until Week 96. Hematology is performed at baseline and days 2, 5, 8, 11, 15, 18, 22, 25 of cycle 1, weekly in cycle 2, then on every scheduled visit (D1 of Cycle 3 to 12, at Cycle 12 Day 28 ,then every 12 weeks) and end of treatment.
Maximum plasma concentration (Cmax) | pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 hours on days 1, 2, and 8
  To characterize the pharmacokinetics (PK) of INC424 alone or in combination with BKM120
Maximum plasma concentration time (Tmax) | pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 hours on days 1, 2, and 8
  To characterize the pharmacokinetics (PK) of INC424 alone or in combination with BKM120
Area under the plasma concentration time curve (AUC) | pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8 hours on days 1, 2, and 8
  To characterize the pharmacokinetics (PK) of INC424 alone or in combination with BKM120
Maximum plasma concentration (Cmax) | pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 24 hours on days 2 and 8
  To characterize the pharmacokinetics (PK) of BKM120 alone or in combination with INC424
Maximum plasma concentration time (Tmax) | pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 24 hours on days 2 and 8
  To characterize the pharmacokinetics (PK) of BKM120 alone or in combination with INC424
Area under the plasma concentration time curve (AUC) | pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 24 hours on days 2 and 8
  To characterize the pharmacokinetics (PK) of BKM120 alone or in combination with INC424
Duration of adverse events | after each cohort is enrolled at baseline until the maximum tolerated dose is established
  Adverse Events are monitored at each study visit and 30 days post last dose of study drug
Severity of adverse events | after each cohort is enrolled at baseline until the maximum tolerated dose is established
  Adverse Events are monitored at each study visit and 30 days post last dose of study drug
Severity of serious adverse events | after each cohort is enrolled at baseline until the maximum tolerated dose is established
  Serious Adverse events monitored at each study visit and 30 days post last dose of study drug
Duration of serious adverse events | after each cohort is enrolled at baseline until the maximum tolerated dose is established
  Adverse Events are monitored at each study visit and 30 days post last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- Australia (2):
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Melbourne, Victoria
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Paris, France
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Rostock
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (2):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Varese, VA
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Madrid, Spain
- United Kingdom (2):
  - Novartis Investigative Site, Edgbaston, Birmingham
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for INC424A2104 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17230